CLINICAL TRIAL: NCT03147157
Title: The Effect of Human Leukocyte Antigen Macthing on Guiding Tacrolimus Regimen
Brief Title: The Effect of Human Leukocyte Antigen Macthing on Guiding Tacrolimus Regimen After Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Guoyue Lv, Vice President, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCPYJJ2017007
Record Dates: First submitted 2017-04-27; First posted 2017-05-10 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Liver Transplantation; Graft Versus Host Disease; Graft Rejection; Drug-Related Side Effects and Adverse Reactions
Keywords: tacrolimus; histocompatibility antigens
MeSH Terms: conditions — Graft vs Host Disease; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- research group,low MR group (Experimental): tacrolimus regimen guided by HLA matching rate
  Interventions: Other: tacrolimus regimen guided by HLA matching rate
- observation group,low MR group (No Intervention): tacrolimus regimen is applied according to clinical experience
- research group,middle MR group (Experimental): tacrolimus regimen guided by HLA matching rate
  Interventions: Other: tacrolimus regimen guided by HLA matching rate
- observation group,middle MR group (No Intervention): tacrolimus regimen is applied according to clinical experience
- research group,high MR group (Experimental): tacrolimus regimen guided by HLA matching rate
  Interventions: Other: tacrolimus regimen guided by HLA matching rate
- observation group,high MR group (No Intervention): tacrolimus regimen is applied according to clinical experience

INTERVENTIONS:
Other: tacrolimus regimen guided by HLA matching rate — required low,middle and high tacrolimus concentration in high,middle and low MR group respectively
  Arms: research group,high MR group; research group,low MR group; research group,middle MR group

SUMMARY:
The aim of this research is to design a randomized controlled clinical study, which is based on HLA matching rate to guide tacrolimus regimen. In this study, the possibility of tacrolimus regimen guided by HLA matching rate will be explored, the occurrence rate of GVHD and rejection reaction will be observed, and the occurrence time and degree of adverse reactions caused by immune inhibitors will be identified. In the meantime, providing a possible prospect for prevention of GVHD and reduction or removal of immune inhibitors.

DETAILED DESCRIPTION:
Liver transplantation is the most effective treatment for end-stage liver disease, yet long term survival is limited by acute and chronic rejection reaction and adverse reactions caused by immune inhibitors. However, effective guideline of immune inhibitors regimen after liver transplantation is lacking. Human major histocompatibility antigens (HLA) is crucial in renal transplantation, while the role in liver transplantation is unclear. It is reported that HLA matching was closely related to the occurrence of graft versus host disease (GVHD) after liver transplantation. And by reducing or removing the immune inhibitors can change the course of illness, improve prognosis, at the same time conduce to induce immune tolerance. Therefore, the investigators have the reason to believe that HLA matching rate has closely association with postoperative immune status of patients after liver transplantation, which may guide immune inhibitors regimen. The aim of this research is to design a randomized controlled clinical study, which is based on HLA matching rate to guide tacrolimus regimen. In this study, the possibility of tacrolimus regimen guided by HLA matching rate will be explored, the occurrence rate of GVHD and rejection reaction will be observed, and the occurrence time and degree of adverse reactions caused by immune inhibitors will be identified. In the meantime, providing a possible prospect for prevention of GVHD and reduction or removal of immune inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* patients signed informed consent，patients with good compliance

Exclusion Criteria:

* autoimmune liver disease,ABO incompatibility,combined organ transplantation,re-transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Possibility of tacrolimus regimen guided by HLA matching rate | 3 months
  Changes of liver function and incidence of acute rejection early after liver transplantation

SECONDARY OUTCOMES:
Occurrence rate of GVHD | 5 years
  Occurrence rate of GVHD between the different groups
Occurrence time of adverse reactions caused by immune inhibitors | 5 years
  Occurrence time of adverse reactions caused by immune inhibitors between the different groups
Degree of adverse reactions caused by immune inhibitors | 5 years
  Degree of adverse reactions caused by immune inhibitors between the different groups
Patient survival rate | 1-year,3-year and 5-year
  Patient survival rate between the different groups